CLINICAL TRIAL: NCT03972241
Title: Three Dimensional Motion Analysis of Daily Activities With Functional Insole in Parkinsonian Patients
Brief Title: Strategy for Daily Activity Improvement in Patients With Parkinson's Disease
Acronym: Parkinson
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kwan-Hwa Lin (Other)
Collaborators: Buddhist Tzu Chi General Hospital (Other)
Responsible Party: Sponsor-Investigator, Kwan-Hwa Lin, Department of Tzu Chi University, Buddhist Tzu Chi General Hospital
Organization: Buddhist Tzu Chi General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB103-43-A; IRB103-42-A (Other: Buddhist Tzu Chi Hospital); IRB 103-173-A (Other: Buddhist Tzu Chi Hospital)
Record Dates: First submitted 2015-01-26; First posted 2019-06-03 (Actual); Last update posted 2019-06-03 (Actual); Status verified 2019-05

CONDITIONS: Parkinson Disease
Keywords: Parkinson disease; Quality of life; Physical therapy; tremor; coordination; gait analysis
MeSH Terms: conditions — Parkinson Disease; Tremor | interventions — Foot Orthoses

STUDY DESIGN:
Intervention Model Description: To compare between experimental and control groups.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): different interventions including foot insole or kinetic training
  Interventions: Device: foot insole
- control (No Intervention): No intervention

INTERVENTIONS:
Device: foot insole — arch support and toe extension
  Other Names: spiral drawing
  Arms: Intervention

SUMMARY:
The symptoms and signs of patients with Parkinson's disease (PD) include bradykinesia, rigidity, tremor and poor sensory integration, which result in mobility disability. Present integrated research project tries to investigate the effects of different physical therapy interventions on daily activities in patients with PD. This integrated research project includes 3 subprojects as follows. The title of Subproject 1 is "Three dimensional motion analysis of daily activities with functional insole in Parkinsonian patients". The title of Subproject 2 is "Immediate and long-term effects of novel plantar mechanical device on postural control in standing and gait performance in people with Parkinson's disease". The title of Subproject 3 is "Upper extremity hand function and coordination during functional movement in patients with Parkinson's disease".

This multidisciplinary research project collaborates with Department of Physical Therapy, and Department of Medicine in Tzu Chi University. Furthermore, this integrated study also works with Department of Neurology, Department of Neurosurgery, as well as Department of Rehabilitation in Tzu Chi Hospital to improve the mobility in patients with PD.

This is a three-year integrated project, and the common purposes of this project in each are as follows. In the first year, it is to compare the daily functional difference between the healthy and the Parkinsonian patients. In the second year, it is to examine the immediate and short-term effects of different interventions on daily activities in Parkinsonian patients.The third year is for upper extremity functional assessment.

DETAILED DESCRIPTION:
In the first year, it is to compare the functional difference of biomechanics and motor control between the healthy and the Parkinsonian patients. In the second year, it is to examine the immediate and short-term effects of functional foot insole and the kinetic training on daily activities in Parkinsonian patients. In the third year, it is to examine the hand tremor during drawing, and the coordination during reaching in Parkinsonian patients.

ELIGIBILITY:
Inclusion Criteria:

* Stage II~IV of Hoehn and Yahr Staging of Parkinson's Disease and normal subjects, whose age between 40~75.

Exclusion Criteria:

* Brain injury or hemorrhage, including stroke, etc.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Ambulation | 1 year
  gait cycle

SECONDARY OUTCOMES:
Foot pressure | 1 year
  center of pressure
Spiral drawing | 1 year
  Figure plot
Coordination | 1 year
  Reaching movement

CONTACTS AND LOCATIONS:
Overall Officials: Kwan-Hwa Lin, PhD, Principal Investigator — Tzu Chi University
Locations (1):
- Tzu Chi University, Hualien City, Hualien County, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yen CY, Lin KH, Hu MH, Wu RM, Lu TW, Lin CH. Effects of virtual reality-augmented balance training on sensory organization and attentional demand for postural control in people with Parkinson disease: a randomized controlled trial. Phys Ther. 2011 Jun;91(6):862-74. doi: 10.2522/ptj.20100050. Epub 2011 Apr 7. PMID 21474638
- [Background] Chen CH, Lin KH, Lu TW, Chai HM, Chen HL, Tang PF, Hu MH. Immediate effect of lateral-wedged insole on stance and ambulation after stroke. Am J Phys Med Rehabil. 2010 Jan;89(1):48-55. doi: 10.1097/PHM.0b013e3181c1ea8a. PMID 19884813
- [Background] Myers KA, Long JT, Klein JP, Wertsch JJ, Janisse D, Harris GF. Biomechanical implications of the negative heel rocker sole shoe: gait kinematics and kinetics. Gait Posture. 2006 Nov;24(3):323-30. doi: 10.1016/j.gaitpost.2005.10.006. Epub 2005 Nov 21. PMID 16300949
- [Background] Morris ME, Huxham F, McGinley J, Dodd K, Iansek R. The biomechanics and motor control of gait in Parkinson disease. Clin Biomech (Bristol). 2001 Jul;16(6):459-70. doi: 10.1016/s0268-0033(01)00035-3. PMID 11427288
- [Background] Lee HJ, Chou LS. Detection of gait instability using the center of mass and center of pressure inclination angles. Arch Phys Med Rehabil. 2006 Apr;87(4):569-75. doi: 10.1016/j.apmr.2005.11.033. PMID 16571399